CLINICAL TRIAL: NCT02792426
Title: A Study to Evaluate the Comparative Pharmacokinetics of Nicotine After Administration Via Research Electronic Nicotine Delivery System S-TA-U001 in Healthy Volunteer Smokers and Current E-Cigarette Users
Brief Title: Nicotine Pharmacokinetics From Research Electronic Nicotine Delivery System S-TA-U001 in Smokers and E-Cigarette Users
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NJOY, Inc. (Industry)
Collaborators: LA Clinical Trials (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: NPK016-N44DA; 271201500019C-0-0-1 (NIH)
Record Dates: First submitted 2016-05-23; First posted 2016-06-07 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Cigarette Smoking
Keywords: Smoking Cessation; Nicotine Dependence; Tobacco Dependence
MeSH Terms: conditions — Cigarette Smoking; Smoking Cessation; Tobacco Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 AB (Active Comparator): Smoker subject's own brand of combustion cigarette
  Interventions: Drug: Research ENDS S-TA-U001; Drug: Nicorette Inhalator
- Group 1 BA (Active Comparator): Smoker subject's own brand of combustion cigarette
  Interventions: Drug: Research ENDS S-TA-U001; Drug: Nicorette Inhalator
- Group 2 (Active Comparator): E-cigarette user's own brand of electronic nicotine delivery system (ENDS)
  Interventions: Drug: Research ENDS S-TA-U001

INTERVENTIONS:
Drug: Research ENDS S-TA-U001
Drug: Nicorette Inhalator
  Arms: Group 1 AB; Group 1 BA

SUMMARY:
To better understand the PK and associated pharmacodynamic (PD) responses produced by the Research ENDS S-TA-U001 product, this study will compare the Research ENDS S-TA-U001 to

* The subject's own brand combustion (non-menthol) cigarette and a U.S. FDA approved smoking cessation product, the NICORETTE Inhalator, in current non-menthol cigarette smokers who have some limited e-cigarette experience (Group 1).
* Commercially available products in current primarily e-cigarette users (experienced ENDS users) (Group 2) The PK/PD session for each product will be conducted in a controlled clinical setting with frequent PK sampling after 14 hours of supervised abstinence from all forms of nicotine. Subjects will familiarize themselves with the Research ENDS S-TA-U001 and NICORETTE Inhalator by using each product in the real world for one day before the PK/PD session for that product.

Primary Objectives:

Group 1 objectives are to characterize the nicotine PK profile (eg, maximum plasma concentration [Cmax], time to maximum plasma concentration [Tmax], area under the concentration-time curve [AUC], and terminal half-life [t1/2]) for 10 inhalation and ad lib sessions of Research ENDS S-TA-U001 and explore how the Cmax compares to a 15 ng/mL level during the 4.5-minute 10 inhalation and the 6 hour ad lib use sessions, to compare the PK profiles between Research ENDS S-TA-U001 to the profiles of combustion cigarettes measured at the baseline session, and to demonstrate superiority of PK profile of Research ENDS S-TA-U001 to that of the marketed NICORETTE Inhalator.

Group 2 objectives are to characterize the nicotine PK profile of Research ENDS S-TA-U001 and explore how the Cmax compares to a 15 ng/mL level during the 4.5-minute 10 inhalation and 6 hour ad lib use sessions, and to compare the PK profile between Research ENDS S-TA-U001 to the profile of a commercial ENDS product measured at the baseline session.

Secondary objectives:

Secondary objectives include comparison of the nicotine PK of the Research ENDS S-TA-U001 to the subjects' normal nicotine source (combustion cigarettes for Group 1 or commercial ENDS for Group 2), to evaluate the safety and tolerability of Research ENDS S-TA-U001, to evaluate the effects on craving and user satisfaction of the Research ENDS S-TA-U001 vs a combustion cigarette or the NICORETTE Inhalator (Group 1) or a commercial ENDS product (Group 2), and to evaluate various biomarkers following use of each test product.

DETAILED DESCRIPTION:
Subjects in Group 1 will participate in a Phase 1 2×2 cross-over study of the Research ENDS S-TA-U001 (Test Product A) and NICORETTE Inhalator (Test Product B). Subjects in Group 2 will participate in a study to examine the effect of the Research ENDS S-TA-U001 (Test Product A).

Approximately 20 healthy volunteers, ages 21 to 65 inclusive, who are current combustion cigarette smokers will be enrolled into Group 1 for the 2×2 cross-over study. Approximately 14 healthy volunteers, ages 21 to 65 inclusive, who are current primarily e cigarette users will be enrolled into Group 2. Initial screening for the study will occur from 7 to 21 days before the first PK assessment/in-clinic device Training Visit on Day 1. Subjects in Group 1 will be randomized to Sequence AB (10 subjects) or Sequence BA (10 subjects).

On Day 1, subjects will arrive at the research site to begin at least 14 hours of overnight supervision to insure abstinence from all forms of nicotine prior to the first administration of the Baseline Product. Each subject will complete a 10 inhalation session of his or her normal nicotine source (either the subject's own brand of a combustion cigarette [Group 1] or the subject's own brand of commercial ENDS product [Group 2]) in 4.5 minutes, abstain for 1 hour 55 minutes, complete a second session of 10 inhalations in 4.5 minutes, complete a 6 hour ad lib use session, and complete a series of behavioral assessments over the PK sampling/observation period lasting 8 hours and 5 minutes. The first series of 4.5-minute 10 inhalation sessions will be videotaped to assess inhalation duration and technique. Subjects will abstain from food for one hour before each 10 puff session and caffeine within one hour of the first 10 puffs through the duration of the entire ad lib session.

Following the sampling/observation period on Day 1, subjects in Group 1 Sequence AB and subjects in Group 2 will be trained on how to properly use the Research ENDS S-TA-U001, and Group 1 Sequence BA subjects will be trained on how to properly use the NICORETTE Inhalator. Prior to discharge, subjects will be provided with two cartridges of the Research ENDS S-TA-U001 or a set of NICORETTE Inhalator for at-home use for 1 day (starting immediately after clinic discharge) depending on the group and sequence to which they are assigned. Subjects will be encouraged (though not required) to use the Research ENDS S-TA-U001 or NICORETTE Inhalator as their exclusive nicotine source. Subjects will record the number of combustible cigarettes smoked (if any) and the number of cartridges of the Research ENDS S-TA-U001 or NICORETTE Inhalator used, depending on sequence (Group 1), or the number of cartridges of the Research ENDS S-TA-U001 used and the amount of e liquid used (if any) from their commercial ENDS products (Group 2). All subjects will be required to return all of the study devices used as well as used and unused cartridges at the next visit.

On Day 3, subjects will arrive at the research site to begin at least 14 hours of overnight supervision to insure abstinence from all forms of nicotine prior to the first administration of the Test Product. Subjects in Group 1 Sequence AB and Group 2 will complete a 10 inhalation session of Research ENDS S-TA-U001 in 4.5 minutes, abstain for 1 hour 55 minutes, complete a second session of 10 inhalations in 4.5 minutes, followed by a 6 hour ad lib use session. Subjects in Group 1 Sequence BA will complete a 10 inhalation session of NICORETTE Inhalator, abstain for 1 hour 55 minutes, complete a second session of 10 inhalations in 4.5 minutes, followed by a 6 hour ad lib use session. A series of behavioral assessments will be performed during the PK sampling/observation period lasting 8 hours and 5 minutes. The first series of 4.5 minute 10 inhalation sessions for both products will be videotaped to assess inhalation duration and technique. Subjects will abstain from food for one hour before each 10 puff session and caffeine within one hour of the first 10 puffs through the duration of the entire ad lib session. Subjects in Group 2 will be discharged from the clinic following the final PK blood draw and completion of all final clinical assessments on Study Day 3. Following the sampling/observation period, subjects in Group 1 Sequence AB will be trained on how to properly use the NICORETTE Inhalator and subjects in Group 1 Sequence BA will be trained on how to properly use the Research ENDS S-TA-U001. Prior to discharge, subjects, depending on the group and sequence to which they are assigned, will be provided with two cartridges of the Research ENDS S TA U001 or a set of NICORETTE Inhalator for at-home use for 1 day (starting immediately after clinic discharge). Subjects will be encouraged (though not required) to use the Research ENDS S-TA-U001 or NICORETTE Inhalator as their exclusive nicotine source. All subjects will be required to return all of the study devices used as well as used and unused cartridges at the next visit.

On Day 5, subjects in Group 1 will arrive at the research site to begin at least 14 hours of overnight supervision to insure abstinence from all forms of nicotine prior to the first administration of the Test Product. Subjects in Group 1 Sequence AB will complete a 10 inhalation session of NICORETTE Inhalator in 4.5 minutes, abstain for 1 hour 55 minutes, complete a second session of 10 inhalations in 4.5 minutes, followed by a 6 hour ad lib use session. Subjects in Group 1 Sequence BA will complete a 10 inhalation session of Research ENDS S-TA-U001 in 4.5 minutes, abstain for 1 hour 55 minutes, complete a second session of 10 inhalations in 4.5 minutes, followed by a 6-hour ad lib use session. A series of behavioral assessments will be performed during the PK sampling/observation period lasting 8 hours and 5 minutes. The first series of 4.5 minute 10 inhalation sessions for both products will be videotaped to assess inhalation duration and technique. Subjects will abstain from food for one hour before each 10 puff session and caffeine within one hour of the first 10 puffs through the duration of the entire ad lib session. Subjects in Group 1 will be discharged from the clinic following the final PK blood draw and completion of all final clinical assessments on Study Day 5.

ELIGIBILITY:
Inclusion Criteria:

For Group 1: in order to participate in the study, potential subjects must:

1. Be males and females of any race between 21 and 65 years of age inclusive
2. Be current combustion cigarette smokers, defined as smoking a minimum of 10 combustion cigarettes per day for a period of at least 3 months, who smoke commercial (non menthol) cigarettes
3. Not be currently planning to quit smoking combustion cigarettes in the next 3 months
4. Have blood cotinine ≥100 ng/mL and carbon monoxide ≥10 ppm at Screening to confirm smoking status
5. Weigh at least 45 kg and have a Body Mass Index (BMI) between 18 and 40 kg/m2, inclusive, at Screening
6. Be healthy, in the Investigator's opinion, according to medical history; physical examination; electrocardiogram (ECG); and clinical chemistry, urine, and hematological laboratory tests
7. Be willing to refrain from using any source of nicotine other than study supplies for the duration of the study confinement period
8. Have vital signs as follows:

   * Resting heart rate between 50 and 90 beats per minute
   * Systolic blood pressure below 150 mm Hg
   * Diastolic blood pressure below 90 mm Hg
9. Have electrolytes (ie, Na, K, Cl, HCO3) and hematocrit that are clinically normal (± 10% of laboratory limits); subjects marginally outside of this range may be eligible at the discretion of the study physician
10. Have liver function tests (ie, total bilirubin, ALT, AST, GGT, and alkaline phosphatase) less than three times the upper normal limit
11. Have kidney function tests (ie, creatinine and BUN) within clinically normal limits (± 10% of laboratory limits) and calculated creatinine clearance > 80 mL/min for females and > 90 mL/min for males
12. Have an ECG performed that demonstrates normal sinus rhythm, normal conductivity, and no clinically significant abnormalities
13. Be able to demonstrate the ability to comply with the inhalation instructions for Test Product administration (Research ENDS S TA U001 and NICORETTE Inhalator), visually confirmed by clinic staff at Screening visit
14. Be able to verbalize understanding of the consent forms, provide written informed consent, and verbalize willingness to comply with the study procedure
15. Have 5-50 days of use of any ENDS product in their life and no use within 7 days before Screening
16. Have no more than 20 days of use of the NICOTROL Inhaler in their life and no use within the 7 days before Screening

For Group 2: in order to participate in the study, potential subjects must:

1. Be males and females between 21 and 65 years of age inclusive
2. Be current daily users of a commercially available ENDS product, with e-liquids of nicotine concentration 10 to 20 mg/mL
3. Consume at least 1 mL per day of e-liquid in their ENDS product
4. Not smoke more than 2 combustion (non menthol) cigarettes per day
5. Have carbon monoxide ≤15 ppm at Screening to confirm limited smoking status
6. Have blood cotinine ≥100 ng/mL at Screening to confirm nicotine dependence
7. Weigh at least 45 kg and have a Body Mass Index (BMI) between 18 and 40 kg/m2, inclusive, at screening
8. Be healthy, in the Investigator's opinion, according to medical history; physical examination; ECG; and clinical chemistry, urine and hematological laboratory tests
9. Be willing to refrain from using any source of nicotine for the duration of the study confinement period
10. Have vital signs as follows:

    * Resting heart rate between 50 and 90 beats per minute
    * Systolic blood pressure below 150 mm Hg
    * Diastolic blood pressure below 90 mm Hg
11. Have electrolytes (ie, Na, K, Cl, HCO3) and hematocrit that are clinically normal (± 10% of laboratory limits); subjects marginally outside of this range may be eligible at the discretion of the study physician
12. Have liver function tests (ie, total bilirubin, ALT, AST, GGT, and alkaline phosphatase) less than three times the upper normal limit
13. Have kidney function tests (ie, creatinine and BUN) within clinically normal limits (± 10% of laboratory limits) and calculated creatinine clearance > 80 mL/min for females and > 90 mL/min for males
14. Have an ECG performed that demonstrates normal sinus rhythm, normal conductivity, and no clinically significant abnormalities
15. Be able to demonstrate the ability to comply with the inhalation instructions for Test Product administration (Research ENDS S TA U001), visually confirmed by clinic staff at Screening visit
16. Be willing to use tobacco-flavored product
17. Be able to verbalize understanding of the consent forms, provide written informed consent, and verbalize willingness to comply with the study procedure

Exclusion Criteria:

For Group 1 and Group 2: in order to participate in the study, potential subjects must not:

1. Have expected inability to comply with study protocol
2. Have used any of the following in the past 30 days: ultra-light, hand or roll-your-own, menthol, or unfiltered combustion cigarettes; any other form of tobacco (eg, chews, dips, pipes, cigars, hookah); or any form of nicotine replacement therapy (eg, patch, gum, lozenge, inhaler, nasal spray).
3. Be pregnant (based on serum test) or nursing (by self-report)
4. Have history or diagnosis of airway disease, including adult onset asthma or chronic obstructive pulmonary disease (including emphysema or chronic bronchitis), use of an inhaler (apart from a nicotine inhaler) in the previous 5 years, or any episodes of wheezing or bronchospasm in the previous 5 years (history of resolved childhood asthma is acceptable)
5. Have baseline spirometry values (FEV1, FVC, and FEV1/FVC) outside of the lower limit of normal as defined by Hankinson et al, Am J Respir Crit Care Med 1999; 159:179-187.
6. Have had treatment with prescription medications within 21 days or over-the-counter medication within 24 hours of the planned first product use occasion, except for oral or hormonal contraceptive therapies.
7. Have used any drugs or substances (except tobacco) known to be strong inducers or inhibitors of any CYP enzymes (formerly known as cytochrome P450 enzymes) within a 28 days period prior to first product administration. For a list of such drugs and substances, please refer to http://medicine.iupui.edu/clinpharm/ddis/main-table/.
8. Have an active cough, recent or chronic, excluding "smoker's cough"
9. Have any active respiratory infection
10. Have a history of clinically significant cardiac, pulmonary, renal, hepatic, endocrine, neurological, gastrointestinal, metabolic, psychiatric, or hematologic disorders
11. Have poor venous access as defined by being unable to draw samples through a catheter at the screening visit
12. Have been hospitalized within 4 weeks before Screening
13. Have received any other investigational treatment or Test Product within 30 days from randomization (or within 5 half-lives of the Test Product, if known, whichever is greater)
14. Have a history of allergic, anaphylactic, or other hypersensitivity reaction to any e cigarette , or any of the components associated with these products such as propylene glycol
15. Have any medical history or condition (including physical) considered by the Principal Investigator and/or admitting physician to place the subjects at increased risk or preclude safe and/or successful completion of the study
16. Have any history of substance abuse, including alcohol abuse within the last 3 months
17. Have a positive result for any drug of abuse (opiates, benzodiazepines, barbiturates or related CNS depressants, amphetamines or related stimulants, or marijuana) at screening or Day -1
18. Be cognitively impaired to a degree that would affect participation. An adequate level of reading and comprehension is needed in order to complete various forms (e.g., behavioural assessments) that are used as dependent variables
19. Have active syphilis (based on the standard confirmatory test (e.g., FTB-abs))
20. Be undergoing HIV treatment with antiviral and non-antiviral therapy or treatment for HIV-related opportunistic infection
21. Do not actively meet the inclusion criteria at the time of screening

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-10-05; Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Nicotine Cmax | ~5 minutes before administration and at 1, 3, 5, 7, 10, 15, 30, 60, 90, 120, 130, 140, 150, 180, 210, 240, 300, 360, 420, and 480 minutes from start of each administration
  Characterize nicotine Cmax of all test products during a 10-puff 4.5-minute session and a 6 hour ad lib use session and compare to a target level of 15 ng/mL
Nicotine AUC | ~5 minutes before administration and at 1, 3, 5, 7, 10, 15, 30, 60, 90, 120, 130, 140, 150, 180, 210, 240, 300, 360, 420, and 480 minutes from start of each administration
  Characterize nicotine AUC from time 0 to the last time point for all test products
Nicotine tmax | ~5 minutes before administration and at 1, 3, 5, 7, 10, 15, 30, 60, 90, 120, 130, 140, 150, 180, 210, 240, 300, 360, 420, and 480 minutes from start of each administration
  Characterize the time when the maximum nicotine concentration is reached for all test products during a 10-puff 4.5-minute session and a 6 hour ad lib use session

SECONDARY OUTCOMES:
Adverse events and vital signs | 5 days
  To evaluate the safety and tolerability of Research ENDS S TA U001 during 4.5-minute 10 inhalation and 6 hour ad lib use sessions. Vital signs include respiratory rate, blood pressure, and oral temperature.
Effects on craving | 5 days
  To evaluate the effects on craving of the Research ENDS S TA U001 versus (vs) a combustion cigarette or the NICORETTE Inhalator (combustion cigarette users) or a commercial ENDS product (e cigarette users). A 5-item Questionnaire of Smoking Urges will be administered at -3, 2.75, 7, 20, 40, 65, 118, 125, 155, 185, 215, 275, 335, 395, and 455 minutes after the first puff of each test product administration.
Effects on user satisfaction | 5 days
  To evaluate the effects on user satisfaction of the Research ENDS S TA U001 versus (vs) a combustion cigarette or the NICORETTE Inhalator (combustion cigarette users) or a commercial ENDS product (e cigarette users). A likeability survey will be administered at the end of the in-clinic session for each test product
White blood cell count | 5 days
  Evaluation of white blood cell count
Carbon monoxide | 5 days
  Evaluation of carbon monoxide in exhaled breath
Spirometry | 5 days
  Evaluation of spirometry

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Nides, PhD, Principal Investigator — LA Clinical Trials
Locations (1):
- LA Clinical Trials, Burbank, California, United States

IPD SHARING:
Plan to Share IPD: Undecided